CLINICAL TRIAL: NCT01498991
Title: Rehabilitation of the Lower Extremity With AMES Following Incomplete Spinal Cord Injury (SCI)
Brief Title: Spinal Cord Injury Leg Rehabilitation
Acronym: AMES
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Shepherd Center, Atlanta GA (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Paul J. Cordo, Study Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007762; R01NS061304-22 (NIH)
Record Dates: First submitted 2011-12-08; First posted 2011-12-26 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injury; Paraplegia; Quadriplegia; Tetraplegia
Keywords: Incomplete Spinal Cord Injury; Rehabilitation; AMES device; Lower Extremity; Gait; Paraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMES Treatment (Experimental): The subject will receive 30 treatment sessions, conducted 3-4 times per week on the AMES device. Each session will consist of testing followed by 40 minutes of treatment time (20 minutes per each leg) using the AMES device.
  Interventions: Device: AMES Treatment

INTERVENTIONS:
Device: AMES Treatment — The AMES device rotates the ankle over a range of 30 degrees while vibrators stimulate the tendons attached to muscles that move the leg. Each participant will receive treatment of both lower extremities. Treatment of the 2 legs will be scheduled to run in the same session. The subject's task is to assist the motion of the device. The AMES treatment device couples assisted movement and tendon vibration (enhanced sensation) in 30 treatments which will each run approximately 40 minutes (20 minutes on the right leg and 20 minutes on the left leg).

SUMMARY:
The purpose of this study is to determine if individuals with incomplete spinal cord injury (SCI) who remain unable to walk normally 1 year after their SCIs are able to sense and move the affected legs better after 10-13 weeks of treatment with a new robotic therapy device.

The hypothesis is that using the AMES device on the legs of chronic subjects with incomplete SCI will result in improved strength, sensation in the legs, and improved functional gait in the treated limbs.

DETAILED DESCRIPTION:
Traumatic spinal cord injury (SCI) affects over 200,000 people in the USA, with several thousand new injuries each year. Most recovery, following SCI, occurs in the six months following surgery. Further recovery after 12 months is unusual.

In this study 10 subjects, more than 1 year post injury, will be enrolled to test the safety and efficacy of a new type of robotic therapy device known as the AMES device. The aim of this Phase I/II study is to investigate the use of assisted movement and enhanced sensation (AMES) technology in the rehabilitation of the legs of participants with incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

* Paraplegia or tetraplegia due to SCI
* At least 1 year post incomplete Spinal Cord Injury
* Can tolerate sitting upright for at least one hour
* Capable of weight-bearing and taking a step with or without an assistive device
* On the ASIA sensory function (light touch), a score of at least 1 at the L4 and L5 level
* Primary ASIA Motor Criterion (PAMC) a total score of 4-12 for hip extensors, knee extensors, ankle dorsiflexors and ankle plantarflexors, with a minimum score of 1 for each of these muscles in the qualifying leg

Exclusion Criteria:

* Fracture of the treated limb resulting in loss of range of motion
* Concomitant TBI or stroke (Patients who sustained mild head injury during the trauma with no evidence of structural abnormalities on brain images will qualify for the study), or other neurological injury or disease
* DVT of the treated extremity
* Peripheral nerve injury of the treated extremity
* Osteo- or rheumatoid-arthritis limiting range of motion
* Contractures equal to or greater than 50% of the normal ROM
* Skin condition not tolerant of device or sitting upright
* Progressive neurodegenerative disorder
* Botox treatment of the treated extremity in the prior 5 month
* Chronic ITB therapy
* Uncontrolled seizure disorder
* Uncontrolled high blood pressure/angina
* Pain in affected limb or exercise intolerance
* Participation in another therapy or activity-based program
* Combined score on ASIA motor function for knee extensors, ankle dorsiflexors and ankle plantarflexors outside the range of 3-9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Cordo, PhD, Study Director — Oregon Health and Science University; Andrew Nemecek, MD, Principal Investigator — Oregon Health and Science University; Deborah Backus, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (2):
- United States (2):
  - Shepherd Center, Crawford Research Center, Atlanta, Georgia
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMES Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AMES Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity
Description: Measured by the GAITRite system
Time Frame: Baseline (pre-treatment), Post-Treatment change from Baseline ( average 13 weeks), 3 months following completion of treatments (average 26 weeks from Baseline).
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Vibration Threshold Test
Time Frame: as for outcome 1
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Modified Ashworth Scale
Time Frame: as for outcome 1
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Timed 10-Meter Walk Test
Time Frame: as for outcome 1
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Gait Assessment Including Step Length and Cadence
Description: Measured by the GAITRite system
Time Frame: as for outcome 1
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Ankle Active Motion Test
Description: The participants will perform an active range-of-motion (ROM) task each time they are treated with the AMES device, in which they move the affected joint to several target joint angles, guided by visual feedback on a display screen on the AMES device.
Time Frame: Prior to each treatment session, on average 3 times a week
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Ankle Strength
Description: The AMES device will test the affected ankle in each direction for maximum strength of voluntary contraction .
Time Frame: Prior to each treatment session, on average 3 times a week
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: ASIA Motor and Sensory Scores for L2-S1
Time Frame: as for outcome 1
Population: The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.
Arm/Group | AMES Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | AMES Treatment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study was not funded and, therefore, enrollment was terminated and the data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes